CLINICAL TRIAL: NCT06810323
Title: The Respiratory Oxygen Adherence Monitor System for COPD With Long Term Oxygen Therapy
Brief Title: The ROAM Research Study Therapy (LTOT) Version
Acronym: ROAM
Status: Recruiting | Type: Observational
Sponsor: University of Virginia (Other)
Collaborators: Barron Associates, Inc. (Industry)
Responsible Party: Principal Investigator, Y. Michael Shim, MD, Professor, Medicine-Pulmonary and Critical Care Medicine, University of Virginia
Other Study IDs: 231682
Record Dates: First submitted 2024-11-15; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this research is to test a device being developed that can see how patients use oxygen therapy over a long period of time. This study will focus on developing a new display part called ROAM module which will be attached to your oxygen source. The display will provide easily-accessible information that can show how you interact with your supplies and the oxygen machine automatically without connecting the oxygen source to the internet or other devices.

DETAILED DESCRIPTION:
The Respiratory Oxygen Adherence Monitor (ROAM) system objectively determines the duration and pattern of adherence to oxygen therapy on a minute-by-minute basis and provides feedback of usage metrics to patients and their clinicians. The purpose of the ROAM monitor is, ultimately, to improve the clinical management of patients with chronic obstructive pulmonary disease (COPD) and patients requiring long-term oxygen therapy (LTOT), to improve health outcomes in these patients, and to reduce costs that arise from the expensive and preventable exacerbations associated with patient non-adherence. The prevalence of COPD poses an enormous burden to the U.S. healthcare system. LTOT is a well-established treatment for patients with oxygen desaturation due to COPD and other cardiopulmonary diseases. The benefits of adequate adherence to LTOT are substantial both to COPD patients (in terms of reduced morbidity and mortality) and to society (in terms of healthcare cost savings). Despite these benefits, patient adherence to LTOT remains poor. The lack of a method to objectively and reliably quantify LTOT usage complicates the challenge of managing these patients. Furthermore, current adherence metrics (e.g., power-on time) fail to provide information regarding the timing of oxygen use within each 24-hour interval. The ROAM system combines several unobtrusive sensing modalities with adaptive algorithms that detect breathing. In this study, the team will develop a patient-ready product prototype targeted at improving patient LTOT adherence.

ELIGIBILITY:
Inclusion Criteria:

Post-Bronchodilator FEV1/FVC <.80

* Race demographics of the recruitment area reflect the population of the Charlottesville Metropolitan Statistical Area (MSA).
* Due to underrepresentation in local demographics, special effort (via targeted advertising) will be made to recruit Hispanic participants to better match national percentages.
* Participants with medical history of COPD
* Subjects has to have a prescription for oxygen use via nasal cannula or mask at home
* At baseline of health with no hospitalization/exacerbation within the past 6 weeks
* Use of Continuous oxygen at baseline

Exclusion Criteria:

Post -Bronchodilator FEV1 < 25%

* Intermittent oxygen use at home
* Inability to understand simple instructions
* No respiratory infections and exacerbation within 6 weeks of study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 100 COPD subjects with continuous oxygen wear
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-01-14 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
In lab validation study to confirm operation of the device | 2 hour
  Repeatability and correlation of the device compared to standard clinical device (pulse ox and heart rate)

SECONDARY OUTCOMES:
Overnight sleep lab testing while wearing the device to correlate the accuracy of the ROAM device using sleep study results. | Overnight ( 8-12 hours)
  Test the performance of the ROAM device overnight.
Long-term ROAM device testing (4 weeks) | 4 weeks
  Testing the ROAM device in an ambulatory setting and follow-up after 2 weeks and return the device after 4 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Yun M Shim, MD, Principal Investigator — Division of Pulmonary and Critical Medicine
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States